CLINICAL TRIAL: NCT05978011
Title: Assessing the Biology of the Injured Lung - Version 1
Brief Title: 2014TP001 - Assessing the Biology of the Injured Lung - Version 1
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2014TP001
Record Dates: First submitted 2023-07-27; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Respiratory Diseases
MeSH Terms: conditions — Respiratory Tract Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Respiratory diseases are very common and are the third leading cause of death in England. As such, there is strong interest in understanding how respiratory disease occurs.

This study intends to understand the changes that occur within diseased/injured lungs obtained from humans. The end goal of this will be to create new drugs to help treat these disorders.

Diseased lungs will be obtained from patients receiving a lung transplant. Lungs will either be placed onto a heart-lung machine, or surgically cut in order to create a model of the lung that can be used experimentally in the laboratory. Using a heart-lung machine, lungs can be maintained outside of the human body for a maximum of 12 hours, allowing the direct assessment of the organ. Using this procedure, we aim to understand the processes that occur within a disease, as well as during repair. Using the model of the lung, we will look at how the body's immune system interacts within a diseased lung.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to provide informed consent
* Patients must be aged between 18-80 years of age

Exclusion Criteria:

-Patients under 16 or over 70 years of age

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Respiratory disorders - lung transplantation
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2014-08-29 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
To identify the mechanisms that occur during lung inflammation, injury and repair and the contribution of immune cells to these processes. | Prior to lung transplantation.
  Cytokines and chemokines within lungs will be assessed to determine inflammatory profiles. This will be done using luminex arrays that allow quantification of a range of immunologic molecules in bronchoalveolar lavage and perfusate samples. This will provide a broad overview of the prevailing local tissue environment. We will also assess this following immunomodulation as this may be significantly altered by the presence of immunomodulatory therapeutics.

SECONDARY OUTCOMES:
Characterise the migration and functional profile of immune cells within the inflamed/damaged lung. | Prior to lung transplantation
  Immune cells obtained from the lungs on the EVLP circuit and cells cultured in the air liquid model will be incubated with antibodies that target specific cellular markers for the detection using flow cytometry. Immune cells can then be characterised and their function determined. The behavioural characteristics and activation status of immune cells will also be determined using flow cytometry, ELISpot/ELISA, immunohistochemistry and qPCR.
Assess the effectiveness of therapeutic agents that can repair lung damage. | Prior to lung transplantation
  Diseased lungs that have been removed from patients during their transplantation will be used as a model to explore novel therapeutic interventions that can modulate inflammation and induce tissue remodelling within the lungs. The entire lungs will be placed within the EVLP circuit and perfused with an acellular solution. Different therapeutic agents will be introduced to the lungs during EVLP and lung function will be monitored. We will determine if lungs have improved via a clinically relevant improvement in lung function (this is the international standard for lung function assessment during EVLP).
Trial therapeutic agents that can modulate the effect of immune cells in response to lung tissue injury. | Prior to lung transplantation
  Diseased lungs that have been removed from patients during their transplantation will be used as a model to explore novel therapeutic interventions that can modulate inflammation and induce tissue remodelling within the lungs. The entire lungs will be placed within the EVLP circuit and perfused with an acellular solution. Different therapeutic agents will be introduced to the lungs during EVLP and lung function will be monitored. We will determine if lungs have improved via a clinically relevant improvement in lung function (this is the international standard for lung function assessment during EVLP).
Identify new therapeutic targets/agents that can reduce the incidence/severity of inflammatory respiratory conditions. | Prior to lung transplantation
  PDiseased lungs that have been removed from patients during their transplantation will be used as a model to explore novel therapeutic interventions that can modulate inflammation and induce tissue remodelling within the lungs. The entire lungs will be placed within the EVLP circuit and perfused with an acellular solution. Different therapeutic agents will be introduced to the lungs during EVLP and lung function will be monitored. We will determine if lungs have improved via a clinically relevant improvement in lung function (this is the international standard for lung function assessment during EVLP).
Cut sections of the lung to culture in an in vitro lung model to assess the effect of various different mechanisms of injury on the function and characteristics of immune cells. | Prior to lung transplantation
  Lungs will be dissected to be used in an in vitro model, generating a morphologically accurate model of the lung. This model will then be used to assess immune cell characteristics.